CLINICAL TRIAL: NCT02180087
Title: Reduce Nonsteroidal Antiinflammatory Drugs Doses for Analgesia After Sternotomy
Acronym: LoDoNSAID
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHU-0198; 2013-003878-27
Record Dates: First submitted 2014-07-01; First posted 2014-07-02 (Estimated); Last update posted 2014-07-02 (Estimated); Status verified 2014-07

CONDITIONS: Cardiac Surgery; Post-operative Pain
Keywords: Cardiac surgery; Post-operative pain; Kétoprofène; Minimum analgesic dose; Morphin consumption; Morphin secondary effects; Patient comfort and satisfaction; Renal fonction
MeSH Terms: conditions — Pain, Postoperative; Personal Satisfaction | interventions — Ketoprofen

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- placebo group (Placebo Comparator): Group 1 : Placebo group (P). 0 mg/kg ketoprofen IV every 6 hours for 48 hours (or 0 mg/kg every 24 hours) for 48 hours
  Interventions: Drug: Ketoprofen
- ketopofen quarter dose (Other): Group 2 : "Ketoprofen quarter dose" (K ¼). 0,125 mg/kg ketoprofen IV every 6 hours (0,5 mg/kg every 24 hours) for 48 hours.
  Interventions: Drug: Ketoprofen
- ketoprofen half-dose (Other): Group 3 : "Ketoprofen half-dose" (K ½). 0,25 mg/kg ketoprofen IV every 6 hours (1 mg/kg every 24 hours) for 48 hours.
  Interventions: Drug: Ketoprofen
- Ketoprofen full dose (Other): Group 4 : "Ketoprofen full dose" (KPD). 0,5 mg/kg ketoprofen IV every 6 hours (or 2 mg/kg every 24 hours) for 48 hours
  Interventions: Drug: Ketoprofen

INTERVENTIONS:
Drug: Ketoprofen

SUMMARY:
Currently, the management of pain after cardiac surgery is based on the concept of multimodal analgesia: Combined use of non-opioid analgesics associated with morphine intravenous analgesia by a system controlled by the patient (patient-controlled analgesia-PCA).

The combination of paracetamol and morphine PCA is very effective on pain at rest, but is limited on pain mobilization and causes the problem of side effects associated with opioid (overdose, sedation, respiratory depression, gastrointestinal intolerance, urinary retention ...) which are contributing factors to increase the length of stay in Intensive Care Unit, an additional cost of care and an increase postoperative morbidity and mortality.

Methods that have proved their effectiveness on pain and mobilization used in postoperative cardiac surgery are: anti-inflammatory drugs (NSAIDs) and / or loco-regional analgesia techniques. NSAIDs enhance analgesia produced by PCA Morphine and allow a reduction in morphine consumption, improved postoperative pain, decreased sedation and decreased postoperative morbidity and mortality.

Adverse effects of NSAIDs are commensurate with their time and exposure dose. Consequently, NSAIDs, in the absence of against-indications, should always be prescribed and used at the lowest effective dose and for the shortest possible time.

Some studies have suggested that lower doses of NSAIDs didn't appear to affect their effectiveness. At present, the investigators have no studies that address the hypothesis from which minimum dose of ketoprofen analgesic effect is obtained.

The investigators hypothesis is that lower dose ketoprofen may have efficacy on pain in the postoperative mobilization of cardiac surgery. The investigators want to find, in their study, this "optimal" ketoprofen dose which would be the minimum dose for clinical efficacy demonstrated dose.

This optimal dose could reduce the number of adverse effects of NSAIDs, but their study will probably not have enough power to prove it. NSAID use at these low doses, in postoperative cardiac surgery, could be extended to patient populations most at risk or for a duration longer than 48 hours.

DETAILED DESCRIPTION:
To answer this hypothesis the investigators will consider starting a study of four groups of patients where appropriate doses to patient weight gradually increasing ketoprofen will be used in seeking the minimum effective dose.

Four groups will be determined by randomization. In all these groups, analgesia will be supplemented by a systematic standard self-administered treatment with morphine and paracetamol.

* Group 1 : Placebo group (P). 0 mg/kg ketoprofen IV every 6 hours for 48 hours (or 0 mg/kg every 24 hours) for 48 hours.
* Group 2 : "Ketoprofen quarter dose" (K ¼). 0,125 mg/kg ketoprofen IV every 6 hours (0,5 mg/kg every 24 hours) for 48 hours.
* Group 3 : "Ketoprofen half-dose" (K ½). 0,25 mg/kg ketoprofen IV every 6 hours (1 mg/kg every 24 hours) for 48 hours.
* Group 4 : "Ketoprofen full dose" (KPD). 0,5 mg/kg ketoprofen IV every 6 hours (or 2 mg/kg every 24 hours) for 48 hours.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for a cardiac surgery (Coronary artery bypass graft, valve replacement)
* Age over 18 years
* Weight between 60 and 100 kg
* Absence of criteria for non-inclusion

Exclusion Criteria:

* Age over 75 years
* Renal insufficiency (MDRD <60 ml / min)
* Hepatic Insufficiency
* Congestive heart failure (EF <40%)
* Insulin-requiring diabetes
* Preoperative coagulation trouble
* History of peptic ulcer or gastrointestinal bleeding
* Allergy to NSAIDs
* Surgery in emergency, aorta surgery, heart transplantation
* Peptic ulcer scalable, history of peptic ulcer or recurrent bleeding (2 or more distinct episodes of bleeding or ulceration objectified)
* Pregnant or lactating women
* Major protected

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-02; Primary Completion 2015-08 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Pain at the mobilization | At the first 48 hours postoperatively
  Pain at the mobilization of the first 48 hours postoperatively, measured every 4 hours by simple numerical scale or VAS (0: no pain to 10: unbearable pain)

SECONDARY OUTCOMES:
Demographic criteria | at day 1
Quantity of sufentanil administered intraoperatively | at day 1
Pain at rest measured by Visual Analogue Scale | at day 1
  Pain at rest measured every 4 hours from H0+4 hours to H+48 hours by Visual Analogue Scale (H0 : sedation stop time, 1 hour before waking)
Total morphine consumption | from H0 to H0+48 hours
Blood gas monitoring 3 times a day | from H0 to H0+48 hours
Time of removal of drains after surgery | at day 1
Resumption of transit characterized by the first gas time after surgery. | at day 1
Nausea occurrence (number of episodes) assessed every 4 hours | from H0 to H0 +48 hours
Vomiting occurrence (number of episodes) assessed every 4 hours | from H0 to H0 +48 hours
Effective Duration of stay in the Intensive Care Unit | at day 1
Patient satisfaction for its first mobilization assessed by simple scale Likert | at H0+ 48 hours
Occurrence of the following complications: Renal respiratory cardiac Neurological infectious Hemorrhagic | From H0 to H0+48 hours
Any readmission to the intensive care unit in the two weeks following the surgery | at day 7

CONTACTS AND LOCATIONS:
Overall Officials: Vedat ELJEZI, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Eljezi V, Biboulet C, Boby H, Schoeffler P, Pereira B, Duale C. The Dose-Dependent Effects of Ketoprofen on Dynamic Pain after Open Heart Surgery. Pain Physician. 2017 Sep;20(6):509-520. PMID 28934782